CLINICAL TRIAL: NCT00899041
Title: In-vivo Study Investigating the Difference in Functional Outcome Between Two Types of Knee Prostheses: the Sigma FB (Depuy, J&J, UK; Standard Implant) and the Sigma RP-F (Depuy, J&J, UK; High-flexion Implant)
Brief Title: Functional Evaluation of a Standard and a High-flexion Knee Prosthesis Using Thigh-calf Contact Force Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Johnson & Johnson Medical BV, The Netherlands (Unknown); Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ORL-FK-08/02
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2011-12

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Prosthesis
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Standard knee prosthesis (Active Comparator): 'standard' knee prosthesis (Sigma FB, J&J, UK).
  Interventions: Procedure: Total Knee Arthroplasty (TKA)
- High flexion knee prosthesis (Active Comparator): 'high flexion' knee prosthesis (Sigma RP-F, J&J, UK).
  Interventions: Procedure: Total Knee Arthroplasty (TKA)

INTERVENTIONS:
Procedure: Total Knee Arthroplasty (TKA) — 28 subjects will receive the standard Sigma FB knee prosthesis. 28 subjects will receive the high flexion Sigma RP-F knee prosthesis.
  Other Names: Sigma RP-F, J&J, UK; Sigma FB, J&J, UK

SUMMARY:
The purpose of this study is to investigate whether subjects receiving a high-flexion knee prosthesis show a better knee function than patients receiving a standard knee prosthesis. Thigh-calf contact force measurements are used to quantify knee function. The investigators' hypothesis is that high-flexion knees show a better knee function.

DETAILED DESCRIPTION:
Study title:

Functional evaluation of a standard and a high-flexion knee prosthesis using thigh-calf contact force measurements.

Objective:

The objective of this study is to investigate whether subjects receiving a high flexion knee prosthesis (Sigma RP-F, J&J, UK) show a better knee function than patients receiving a standard knee prosthesis (Sigma FB, J&J, UK).

Study Design:

Prospective double blind randomized study.

Study population:

Subjects who will receive total knee arthroplasty (TKA) because of invalidating gonarthritis based on primary osteoarthritis or rheumatic disorders or trauma.

Intervention:

* 28 subjects will receive the standard Sigma FB knee prosthesis.
* 28 subjects will receive the high flexion Sigma RP-F knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving a total knee replacement due to disabling gonarthrosis (cartilage damage):

* Primary due to osteo-arthritis
* Secondary due to rheumatoid arthritis or trauma

Exclusion Criteria:

* Patients suffering from juvenile rheuma
* Patients suffering from hemophilia
* Patients that are incapable to give informed consent
* Patients who receive a total knee replacement due to an oncological resection
* Patients who have received a total knee replacement on the contralateral leg
* Patients who have disabling gonarthrosis on both legs
* Patients having a BMI < 25 kg/m^2
* Patients who have to receive a different prosthesis than used in this study for biomechanical reasons (e.g. revision prosthesis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Thigh-calf contact force | pre-op and 1-year post-op

SECONDARY OUTCOMES:
Passive/active maximal knee flexion angle | pre-op and 1-year post-op
BMI, weight and length | pre-op and 1-year post-op
Thigh and calf circumference | pre-op and 1-year post-op
IKS, WOMAC and VAS (pain/satisfaction) score | pre-op and 1-year post-op

CONTACTS AND LOCATIONS:
Overall Officials: Nico Verdonschot, Prof., Principal Investigator — Radboud University Medical Center
Locations (1):
- Canisius-Wilhelmina Hospital, Nijmegen, Netherlands

REFERENCES:
- [Background] Zelle J, Barink M, Loeffen R, De Waal Malefijt M, Verdonschot N. Thigh-calf contact force measurements in deep knee flexion. Clin Biomech (Bristol). 2007 Aug;22(7):821-6. doi: 10.1016/j.clinbiomech.2007.03.009. Epub 2007 May 18. PMID 17512647
- [Derived] van der Ven PJP, van de Groes S, Zelle J, Koeter S, Hannink G, Verdonschot N. Kneeling and standing up from a chair as performance-based tests to evaluate knee function in the high-flexion range: a randomized controlled trial comparing a conventional and a high-flexion TKA design. BMC Musculoskelet Disord. 2017 Aug 1;18(1):324. doi: 10.1186/s12891-017-1657-3. PMID 28764691